CLINICAL TRIAL: NCT05181982
Title: Wissenschaftliche Evaluation Des Modellvorhabens (§ 64b SGB V) am Pfalzklinikum (EVA_Pfalz)
Brief Title: Evaluation of a Flexible and Integrative Psychiatric Care Model at the Pfalzklinikum (EVA_Pfalz)
Acronym: EVA_Pfalz
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: ISMG, Medical Faculty, Otto-von-Guericke University Magdeburg (Unknown); Scientific Institute for Health Economics and Health System Research, Leipzig (WIG2) (Unknown)
Responsible Party: Principal Investigator, Anne Neumann, Principle Investigator, Head of Mental Health Services Research, PhD, Technische Universität Dresden
Other Study IDs: EVA_Pfalz
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Care
Keywords: Cross-sectoral Treatment; Flexible and Integrated Treatment; Global Treatment Budget; FIT; Psychiatry; Evaluation; Claims data; Cohort study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention Group: Patients being treated at the FIT hospital (Pfalzklinikum) between January 2020 and December 2023
  Interventions: Other: FIT contract with global treatment budget
- Control group: Patients being treated in standard care (control hospitals) in the German federal state Rheinland-Pfalz

INTERVENTIONS:
Other: FIT contract with global treatment budget — Several SHI funds have established a contract (duration = at least eight year) with the model hospital for an alternative remuneration / financing of patients treated in the model hospital (FIT hospital, Pfalzklinikum). This contract encourages the model hospital an alternative treatment of their patients (insured with the involved SHI funds), for example fewer inpatient and more outpatient treatment. The contract is based on a global treatment budget (pre-defined fix budget for a specified number of patients independent from the setting of treatment in the hospital).
  Groups: Intervention Group

SUMMARY:
This study is an evaluation of the flexible and integrative psychiatric care model (according to § 64b of the German Social Code Book V (SGB V)) (FIT) at the Pfalzklinikum. The central concern of this evaluation is to answer the question whether the FIT model offer advantages over standard care. The orientation of model care is a more cross-sectoral provision of services through more flexible treatment intensities.

DETAILED DESCRIPTION:
The introduction of Section 64b SGB V created the possibility of agreeing so-called FIT model projects for the further development of care for mentally ill people. The objective is to improve cross-sectoral care or optimize patient care. More than 20 statutory health insurance (SHI) funds have developed a FIT model project at the Pfalzklinikum in Germany targeting children, youth and adults. By now, this is the largest FIT project within Germany and the only one in the German Federal State Rheinland-Pfalz. There are more 22 FIT projects at German psychiatric hospitals by December 2021. This FIT project started on 01 January 2020 with an initial duration of eight years.

The goal of the contract is the implementation and further development of improved patient care within the framework of a global treatment budget. To optimize care, "Assertive Community Treatment (ACT)" was introduced as treatment in the patient's environment (home). ACT aims to strengthen patient care, especially in outreach treatment (home treatment), and gives treatment providers more flexibility to adapt the type, duration and intensity of treatment to the patient's needs. Furthermore, the model project aims at a continuous treatment and stabilization of the patients in consideration of their social and professional environment, the creation of a continuity of treatment, the increase of the acceptance of the patient-oriented, psychotherapeutic and sociotherapeutic interventions. Furthermore, the change in financing in the form of a global treatment budget should lead to a more effective use of financial resources.

In accordance with § 65 SGB V, all model projects under § 64b SGB V, must be scientifically evaluated by an independent expert (expert team). Eighteen of the 22 FIT projects are under evaluation with a similar study design elsewhere (Neumann et al., 2018), while for the evaluation of another FIT project a slightly adopted design with a multi-methods approach is used (Neumann et al., 2021). The aim of this evaluation is to examine the achievement of the objectives of the FIT model project based on anonymized claims data (March et al, 2020). The main goals of the model project are to shorten the duration of inpatient stays while intensifying day care and / or outpatient forms of treatment, decrease sick leave days, increase treatment continuity, reduce inpatient readmission rate and not to deteriorate further disease- and care-related aspects, such as disease progression or comorbidities. In addition, the total costs of the FIT model care should not exceed those of the standard care or, at a maximum of the same costs, better results should be achieved. However, it is expected that some costs will increase (e.g. outpatient care) while other costs will decrease (e.g. inpatient care) .

The effectiveness, costs, and cost-effectiveness of the FIT model hospital compared to standard care are to be examined. The study presented here is a controlled cohort study utilizing anonymous claims data. The controlled design is based on the fact that information of patients from the intervention hospital, the Pfalzklinikum, is compared to information of comparable patients from structurally similar psychiatric hospitals in the same federal state (Petzold et al, 2019).

ELIGIBILITY:
Inclusion Criteria:

* treatment at the Pfalzklinikum or control hospital after 01.01.2020 (date included) and before 31.12.2023 (date included) with one of the following diagnoses as main diagnosis (ICD-10: F00, F01, F02, F03, F07, F10, F20-29, F30-39, F43, F45, F40-48, F50, F60.31, F70-79, F84, F90-F98, B22 & F02.8, G20.0 & F02.3, G30.0 & F00.0, G30.1 & F00.1) at the department of psychiatry (FA 29xx), department of child and adolescent psychiatry (F30xx) or department of psychosomatic/psychotherapy (FA31xx)
* being insured with any of the participating SHI funds

Exclusion Criteria:

* less than one year follow-up data available
* non-permanent residence in Germany during observation period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anonymized data of the participating SHI funds will be analyzed. This includes all patients being treated at the Pfalzklinikum or a control hospital between 01 January 2020 and 31 December 2023 using claims data up to 31 December 2024 enabling an individual follow-up period of at least 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Duration of inpatient psychiatric treatment | one year prior to recruitment compared to first to fourth year after recruitment
  Days with inpatient stays of each included patient will be marked within the patient-individual follow-up period. A billing matrix defining the type of charge and describing the count will be used to mark days with inpatient stays. Inpatient stays that range outside the patient-specific follow-up time will be censored. The proportion of patients with at least one inpatient stay will be presented. Furthermore, the days of inpatient stays per patient will be added, including the stay that led to inclusion in the evaluation. The classification into inpatient and day care is based on the corresponding charges. If inpatient and day care cases are billed on one day in one hospital, this day will be counted as an inpatient day. It will be analyzed how long patients were treated in hospitals (here only inpatient stays), summed over the entire observation period for each case (all patients).
Sick leave days | one year prior to recruitment compared to first to fourth year after recruitment
  The number of sick leave days due to any mental disorder among employed persons will be counted.

SECONDARY OUTCOMES:
Duration of day care psychiatric treatment | one year prior to recruitment compared to first to fourth year after recruitment
  Days with day care stays of each included patient will be marked within the patient-individual follow-up period. A billing matrix defining the type of charge and describing the count will be used to mark days with day care stays. Day care stays that range outside the patient-specific follow-up time will be censored. The proportion of patients with at least one day care stay will be presented. Furthermore, the days of day care stays per patient will be added, including the stay that led to inclusion in the evaluation. The classification into inpatient and day care is based on the corresponding charges. If inpatient and day care cases are billed on one day in one hospital, this day will be counted as an inpatient day. It will be analyzed how long patients were treated in hospitals (here only day care stays), summed over the entire observation period for each case (all patients).
Outpatient psychiatric treatment in the hospital | one year prior to recruitment compared to first to fourth year after recruitment
  The number of days with a contact in the psychiatric outpatients departments (PIA) in the IG and CG will be recorded and compared. The annual and cumulative number of PIA contacts will be determined on the basis of the PIA documentation.
Effects of special services | one year prior to recruitment compared to first to fourth year after recruitment
  Patients with ACT treatment in the IG will be described in more detail in regard to readmission rate and total costs. Sub-analyses regarding the influence of special services will be conducted and a joint conclusion will be drawn on the effects of special services.
Prevention of treatment discontinuation | one year prior to recruitment compared to first to fourth year after recruitment
  The number of patients with contact to the outpatient section within 30 and 90 days after hospital discharge, the frequency of severely mentally ill patients with no contact to the psychiatric care system within 180 days and the percentage of patients with more than three different service providers within the same care sector will be investigated.
Inpatient hospital readmission | first year after first full inpatient psychiatric discharge after recruitment
  The proportion of persons with an inpatient stay who were readmitted as inpatients within one year after discharge from the hospital and the days between first inpatient discharge and second inpatient treatment will be examined. The follow-up period is determined on a patient-specific basis. For this purpose, the first discharge date from an inpatient stay in the reference hospital (IG or CG) after inclusion into the evaluation that allowed a one-year follow-up period will be taken as the basis. Readmission is given if the patient had a psychiatric diagnosis (ICD-10: Fx) as main diagnosis and was readmitted with a psychiatric diagnosis as main diagnosis within one year.
Further disease- and care-related aspects: comorbidities | one year prior to recruitment compared to first to fourth year after recruitment
  The number of comorbidities will be determined for each patient within the follow-up period and compared between IG and CG. Comorbidities are defined based on the diagnoses of the Elixhauser Score, the diagnosis groups are added unweighted in the context of this analysis.
Further disease- and care-related aspects: mortality | one year prior to recruitment compared to first to fourth year after recruitment
  The proportion of individuals who die within a defined period of time after inclusion in the evaluation will be analyzed and compared.
Further disease- and care-related aspects: disease progression | one year prior to recruitment compared to first to fourth year after recruitment
  The proportion of patient who transition from F32.0 or F32.1 (mild/moderate depressive episode) to F32.2 or F32.3 (severe depressive episode) or from F32 (depressive episode) to F33 (recurrent depressive disorder) or from no addictive disorder (F10-F19) to any additive disorder (F10-F19) will be recorded and compared.
Further disease- and care-related aspects: guideline adherence | one year prior to recruitment compared to first to fourth year after recruitment
  Quality indicators for alcohol dependence, dementia, depression and schizophrenia according to Großimlinghaus et al (2013) which can be mapped with claims data will be examined.
Further disease- and care-related aspects: continuity of care | one year prior to recruitment compared to first to fourth year after recruitment
  It will be analyzed how many cases had at least one contact with the outpatient sector after hospital discharge. A distinction will be made between the outpatient sector in the hospital (PIA) and the outpatient sector outside the hospital (contracted medical sector). In addition, the area of continuity of treatment in the "psychiatric sector" (PIA, physician for psychiatry or child and adolescent psychiatry or psychotherapist) will be summarized.
Direct medical care costs | one year prior to recruitment compared to first to fourth year after recruitment
  The difference in the costs for the treatment of mental illnesses arising between IG and CG during the observation period will be analyzed. In addition, somatic costs will be estimated. For this purpose, the care costs of the following areas will be taken into account: costs of inpatient and day care, cost of outpatient care in hospitals, costs of SHI-accredited medical care, drug costs and remedies costs.
Cost-effectiveness (direct medical costs) | one year prior to recruitment compared to first to fourth year after recruitment
  To compare the efficiency of the model project with standard care, a cost-effectiveness analysis will be performed taking a SHI-funds perspective. The incremental cost-effectiveness ratio will be determined using the primary outcome parameter cumulative duration of inpatient stays as the effect measure.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Neumann, Dr., Study Chair — Center For Evidence-Based Healthcare (ZEGV), Technische Universität Dresden, Germany
Locations (1):
- Center For Evidence-Based Healthcare, Technische Universität Dresden, Dresden, Germany

REFERENCES:
- [Background] Grossimlinghaus I, Falkai P, Gaebel W, Janssen B, Reich-Erkelenz D, Wobrock T, Zielasek J. [Developmental process of DGPPN quality indicators]. Nervenarzt. 2013 Mar;84(3):350-65. doi: 10.1007/s00115-012-3705-4. German. PMID 23494246
- [Background] Quan H, Sundararajan V, Halfon P, Fong A, Burnand B, Luthi JC, Saunders LD, Beck CA, Feasby TE, Ghali WA. Coding algorithms for defining comorbidities in ICD-9-CM and ICD-10 administrative data. Med Care. 2005 Nov;43(11):1130-9. doi: 10.1097/01.mlr.0000182534.19832.83. PMID 16224307
- [Background] Petzold T, Neumann A, Seifert M, Kuster D, Pfennig A, Weiss J, Hackl D, Swart E, Schmitt J. [Identification of Control Hospitals for the Implementation of the Nationwide and Standardized Evaluation of Model Projects According to section sign 64b SGB V: Analysis of Data from Structured Quality Reports]. Gesundheitswesen. 2019 Jan;81(1):63-71. doi: 10.1055/s-0042-116436. Epub 2016 Nov 15. German. PMID 27846670
- [Background] March S, Zimmermann L, Kubat D, Neumann A, Schmitt J, Baum F, Schoffer O, Arnold K, Seifert M, Kliemt R, Hackl D, Pfennig A, Swart E. [Methodological Challenges when Using Claims Data of more than 70 Statutory Health Insurances - A Progress Report from the EVA64 Study]. Gesundheitswesen. 2020 Mar;82(S 01):S4-S12. doi: 10.1055/a-1036-6364. Epub 2020 Jan 21. German. PMID 31962364
- [Background] Neumann A, Swart E, Hackl D, Kliemt R, March S, Kuster D, Arnold K, Petzold T, Baum F, Seifert M, Weiss J, Pfennig A, Schmitt J. The influence of cross-sectoral treatment models on patients with mental disorders in Germany: study protocol of a nationwide long-term evaluation study (EVA64). BMC Psychiatry. 2018 May 18;18(1):139. doi: 10.1186/s12888-018-1721-z. PMID 29776348
- [Background] Neumann A, Hense H, Baum F, Kliemt R, Seifert M, Harst L, Kubat D, Maicher B, Schrey C, Schmitt J, Pfennig A, Weinhold I, Swart E, Soltmann B. Evaluation of a flexible and integrative psychiatric care model in a department of child and adolescent psychiatry in Tubingen, Germany: study protocol (EVA_TIBAS). BMC Health Serv Res. 2021 Nov 22;21(1):1262. doi: 10.1186/s12913-021-07226-1. PMID 34802427